CLINICAL TRIAL: NCT04499690
Title: Managing Cancer and Living Meaningfully (CALM): A Global Initiative
Brief Title: Global CALM Implementation Study
Acronym: Global CALM
Status: Terminated | Type: Observational
Why Stopped: Study recruitment & data collection ceased in Dec 2022 in part due to funding shortages and the impact of the COVID-19 Pandemic. 40 clinician-participants consented; 35 completed measures; no data were analyzed or published; REB was closed Nov 2024.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 18-5670
Record Dates: First submitted 2020-07-24; First posted 2020-08-05 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Depression
Keywords: Psychosocial; Behavioural Intervention; Implementation Science
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Global CALM Training Program Clinicians: Clinicians engaging in the CALM Training Program.
  Interventions: Behavioral: Managing Cancer and Living Meaningfully

INTERVENTIONS:
Behavioral: Managing Cancer and Living Meaningfully — A brief, individual, manualized psychosocial intervention for patients with advanced and metastatic cancer

SUMMARY:
This study seeks to evaluate the implementation of the Managing Cancer and Living Meaningfully (CALM) Program in diverse cultural settings, including its feasibility, fidelity, and acceptability. It will also assess the cross-cultural generalizability of the CALM intervention with a particular focus on patient-reported outcomes with regard to psychological well-being and quality of life.

DETAILED DESCRIPTION:
CALM is a semi-structured, manualized, individual psychotherapy designed for patients with advanced cancer and their loved ones. Research conducted over the past decade has shown that CALM is a feasible, acceptable, and effective therapy for patients with advanced or metastatic cancer.

The CALM Training Program was developed to train oncology clinicians in the delivery of CALM. The training program consists of: 1) introductory workshops, which provide foundational training in the intervention; 2) advanced workshops, which support the development of advanced therapeutic skills; and 3) ongoing case supervision, delivered in small-group format, either in-person or online, which provides an opportunity for continuing improvement and refinement in the delivery of CALM.

To evaluate the implementation of the CALM Program at the clinician and organization levels, we will approach clinicians engaging in the CALM Training Program and invite them to participate in this research study, which includes completion of quantitative measures at baseline, 1 year (primary endpoint) and 2 years (study endpoint), participation in qualitative interviews, and collection of feasibility data. Implementation science frameworks will be applied to assess participants' perceived individual- and contextual-level barriers and facilitators to implementing CALM through qualitative interviews.

Sites involved in the Global CALM Program will conduct pilot studies of CALM in their setting to evaluate CALM at the patient- and caregiver-levels. We will not be involved in the collection of prospective patient- and caregiver-level data, however data will be pooled and analyzed to assess the cross-cultural generalizability of the CALM intervention.

ELIGIBILITY:
Inclusion Criteria:

The research team will approach clinicians who:

* have expressed interest in taking part in the Global CALM Program;
* able to deliver psychotherapeutic care according to the legislation/organizational policy that regulates their profession;
* ≥18 years of age;
* able to provide informed consent;
* fluent in English (or other language(s) in which training and supervision will be offered);
* fluent in the main language spoken in the country where their centre is located (to be able to deliver CALM sessions); and
* willing/able to engage with training in the CALM therapy and attend in-person or online supervision meetings (based on feasibility).

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinicians who are participating in the Global CALM Training Program.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Change in Site Feasibility Metrics | Throughout study completion, every 12 months
  The Global CALM Program's site lead will complete site feasibility metrics, which include measures of reach (e.g. # clinicians engaged in CALM training, # of CALM-related research projects), effectiveness (e.g. CALM treatment integrity and supervision evaluation ratings), adoption (e.g. # of patients being seen for CALM), implementation (e.g. # of completed CALM cases, # CALM certified therapists), and maintenance. This measure is completed annually throughout the site's engagement in the CALM Program.
Change in Confidence in Therapy - Oncology Questionnaire | Changes from baseline, 1 Year, and 2 Years
  The Confidence with Therapy - Oncology Questionnaire (CTO) is a 14-item Likert-type questionnaire used to assess a therapists' level of confidence in the delivery of psychotherapy to patients who are living with advanced cancer. This questionnaire will be administered to participating clinicians who partake in case supervision, at baseline, 1 year, and 2 years.
Change in Supervision Evaluation Questionnaire | Changes from baseline, 1 Year and 2 Years
  The CALM Supervision Evaluation Questionnaire is a 30-item questionnaire evaluating CALM supervision meetings. Adapted from the works of Spiegel and Spira (1991), Arcinue (2002), Winstanley (2000), and Cliffe et al. (2016), this questionnaire evaluates the perceived feasibility, acceptability and efficacy of supervision, the extent to which the supervision adhered to CALM therapy protocol, and the overall experience of participating in group supervision. This questionnaire will be administered to clinicians who partake in case supervision, at the 1- and 2-year time points.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Rodin, MD, Principal Investigator — University Health Network, Toronto; Sarah Hales, MD PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada